CLINICAL TRIAL: NCT04509050
Title: A Prospective Study to Evaluate Biological and Clinical Effects of Significantly Corrected CFTR Function in Infants and Young Children (BEGIN Study)
Brief Title: Study to Evaluate Biological & Clinical Effects of Significantly Corrected CFTR Function in Infants & Young Children
Acronym: BEGIN
Status: Recruiting | Type: Observational
Sponsor: Sonya Heltshe (Other)
Collaborators: Cystic Fibrosis Foundation (Other); University of Washington (Other); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor-Investigator, Sonya Heltshe, Associate Professor University of Washington, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Other Study IDs: BEGIN-OB-19
Record Dates: First submitted 2020-08-06; First posted 2020-08-11 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; CF; CFTR Modulator; triple combination therapy; elexacaftor; tezacaftor; ivacaftor
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; ivacaftor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma, Buffy Coat, Urine, Stool, oropharyngeal (OP) swab, Bronchoalveolar lavage (BAL)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Part A: Children with CF not on ivacaftor or elexacaftor/tezacaftor/ivacaftor CFTR modulator therapy.
- Part B: Children with CF planning to start ivacaftor or elexacaftor/tezacaftor/ivacaftor CFTR modulator therapy. Participants from the Part A cohort of this study may enroll into the Part B cohort if they become eligible for these CFTR modulator therapies and plan to start them.
  Interventions: Drug: Ivacaftor or elexacaftor/tezacaftor/ivacaftor

INTERVENTIONS:
Drug: Ivacaftor or elexacaftor/tezacaftor/ivacaftor — In Part B, approved CFTR modulator as prescribed at the discretion of the treating physician -not dictated by the BEGIN investigators
  Other Names: Kalydeco or Trikafta; Vertex (VX)-770 or VX-445/VX-661/VX-770
  Groups: Part B

SUMMARY:
This is a two-part, multi-center, prospective longitudinal, exploratory study of highly effective cystic fibrosis transmembrane conductance regulator (CFTR) modulators and their impact on children with cystic fibrosis (CF).

DETAILED DESCRIPTION:
This is a two-part, multi-center, prospective longitudinal, exploratory study of highly effective cystic fibrosis transmembrane conductance regulator (CFTR) modulators and their impact in children with cystic fibrosis (CF) on endocrine growth factors and height, gastrointestinal function and gut microbiome, lung function and respiratory microbiome, liver and pancreatic function, sweat chloride, inflammatory markers, and bone health.

Total duration of the study is expected to be 10 years. Part A will be a prospective cross-sequential study to describe the natural history of hormonal growth factors in early childhood and assess the feasibility of additional measurements. In Part A, subjects will have up to 8 visits over a period of up to 5 years.

Part B will be a prospective longitudinal study to observe the effects of administration of either ivacaftor or elexacaftor/tezacaftor/ivacaftor (elex/tez/iva) on growth. In Part B, subjects will have 1 "before ivacaftor or elex/tez/iva" visit within 30 days before initiation of the therapy and 8 "after ivacaftor or elex/tez/iva" visits over a 60-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Part A:

  * Less than 10 years of age at the first study visit.
  * Documentation of a CF diagnosis.

Part B:

* Participated in Part A OR less than 7 years of age at the first study visit.
* Documentation of a CF diagnosis.
* CFTR mutations consistent with FDA labeled indication of highly effective modulator therapy (ivacaftor or elexacaftor/tezacaftor/ivacaftor).
* Physician intent to prescribe ivacaftor or elexacaftor/tezacaftor/ivacaftor.

Exclusion Criteria:

* Part A and Part B:
* Use of an investigational drug within 28 days prior to and including the first study visit.
* Use of ivacaftor or elexacaftor/tezacaftor/ivacaftor within the 28 days prior to and including the first study visit.
* Use of chronic oral corticosteroids within the 28 days prior to and including the first study visit.

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Part A - children with confirmed diagnosis of cystic fibrosis who are less than 10 years of age and not on ivacaftor or elexacaftor/tezacaftor/ivacaftor CFTR modulator therapy
  Part B - children with confirmed diagnosis of cystic fibrosis who are less than 7 years of age (or participated in Part A of the study) with an intention to start ivacaftor or elexacaftor/tezacaftor/ivacaftor CFTR modulator therapy
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Part A Primary Outcome Measure: Change in weight-for-age z-scores | Baseline to 12 months
  Weight-for-age z-scores over time
Part A Primary Outcome Measure: Change in height-for-age z-scores | Baseline to 12 months
  Height-for-age z-scores over time
Part B Primary Outcome Measure: Change in weight-for-age z-scores | Baseline to 12 months
  Change in weight-for-age z-scores from baseline
Part B Primary Outcome Measure: Change in height-for-age z-scores | Baseline to 12 months
  Change in height-for-age z-scores from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Ramsey, MD, Principal Investigator — Seattle Children's Hospital; Lucas Hoffman, MD PhD, Principal Investigator — University of Washington/Seattle Children's; Katie Larson Ode, MD, Principal Investigator — University of Iowa
Locations (35):
- United States (35):
  - The Children's Hospital Alabama, University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University Medical Center, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - The Nemours Children's Clinic - Orlando, Orlando, Florida
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Michigan Medicine, Ann Arbor, Michigan
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - The Minnesota Cystic Fibrosis Center, Minneapolis, Minnesota
  - Children's Mercy Kansas City, Kansas City, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - The Cystic Fibrosis Center of Western New York, Buffalo, New York
  - Children's Hospital of New York, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - New York Medical College at Westchester Medical Center, Valhalla, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oklahoma Cystic Fibrosis Center, Oklahoma City, Oklahoma
  - Oregon Health Sciences University, Portland, Oregon
  - Hershey Medical Center Pennsylvania State University, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - University of Texas Southwestern / Children's Health, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Primary Children's Cystic Fibrosis Center, Salt Lake City, Utah
  - Vermont Children's Hospital, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No